CLINICAL TRIAL: NCT06829706
Title: A Randomized Trail Protocol to Access Efficacy of Modified Olfactory Training Method for Patients With Post-viral Olfactory Dysfunction
Brief Title: The Efficacy of Modified Olfactory Training Method for Patients With Post-viral Olfactory Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9059103
Record Dates: First submitted 2025-02-06; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Olfactory Dysfunction; Post Viral Olfactory Dysfunction (PVOD)
Keywords: Olfactory Training; Modified Olfactory Training Device; Post Viral Olfactory Dysfunction (PVOD)

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Conventional olfactory training (Active Comparator): Patients allocated to the COT group are told to expose themselves twice daily to four odors (phenyl ethyl alcohol: rose, menthol: mint, citronellal: lemon, and eugenol: cloves)，which are placed in four brown glass jars (total volume 50 mL) with one of the four odors in each (1 mL each, soaked in cotton pads to prevent spilling). All jars are labeled with the odor name.
  Olfactory training includes exposure to odorants twice per day for 5 minutes. Every olfactory session included rotated exposure to each odorant for 10 seconds each, with time intervals of 10 seconds between odors. The resting order of the four odors is mint-rose-lemon-clove.
  Patients were advised to sniff the odors in the morning before breakfast and in the evening before bedtime.
  Interventions: Device: Conventional olfactory training device
- The Control group (Sham Comparator): The COT group will differ solely with regard to the ingredients contained in the training jars given to the participants. Whereas in the COT group, the training jars will contain the active odors previously selected, in the placebo group, the training jars will be filled with a placebo odorless solvent (propylene glycol). To increase the overall compliance and to ascertain that the placebo (odorless) group remains blinded to the treatment allocation, all patients are told that whereas the odors used during the therapy tend to be less strong, and may be insufficiently intense to produce an odor sensation (i.e., subliminal odors), they are intense enough to be perceived by the brain and may influence mental processes and behavior. The training will last for 12 weeks. After the study completion, all participants will be individually contacted and their group allocations will be revealed. All patients will be offered the possibility of performing or continuing a training with odors.
  Interventions: Device: Conventional olfactory training device with placebo
- The Modified olfactory training (Experimental): When the patient is doing olfactory training, he/she selects an odor and installs the corresponding odor bottle on the new olfactory training device. Insert the nose end into one nostril, hold the mouth end in the mouth, take a deep breath through the nose, blow out slowly for about 7 seconds, and carefully experience the changes in the nature and intensity of the nasal odor. Immediately remove the device from the nostril and mouth, take a slow, natural breath through the nose for about 3 seconds; Repeat the above operation for a total of three cycles. The operation steps for the other nostril are the same as those above. When both nostrils have finished sniffing the same odor, stop the training, breathe freely, and rest for 10 seconds. Then continue to sniff the next odor and train in the order and method described above.
  Accordingly, all odors used for the application of MOT were identical to the COT method in terms of the duration and application time of each session.
  Interventions: Device: Modified olfactory training device

INTERVENTIONS:
Device: Conventional olfactory training device — Conventional olfactory training was designed by Hummel et al. They performed OT using four odors (phenyl ethyl alcohol, rose; eucalyptol, eucalyptus; citronella, lemon; and eugenol, cloves), which are representative of four odor categories on the odor prism proposed by Henning.
  Arms: The Conventional olfactory training
Device: Modified olfactory training device — Participants will use a modified olfactory training device based on expiratory pressure. Its bidirectional airflow and unidirectional pressure characteristics significantly increased the deposition rate of olfactory odors in the olfactory cleft area, making the patient feel stronger in the nasal cavity during olfactory training.
  Arms: The Modified olfactory training
Device: Conventional olfactory training device with placebo — Based on the traditional olfactory training device, four olfactory odors are replaced by placebo。
  Arms: The Control group

SUMMARY:
The goal of this clinical trial is to validate the effectiveness of the modified olfactory training device, the main questions it aims to answer are: Is the modified olfactory training device effective in treating patients with post-viral olfactory dysfunction? Compared to the conventional device, how efficient is the modified olfactory training device for improving olfactory function?

DETAILED DESCRIPTION:
Background The aim of this article is to present the research protocol for a randomized, controlled, multi-center, placebo study that will assess the olfactory function and the effect of an intervention based on olfactory training in patients with post-viral olfactory dysfunction, and compare it with traditional olfactory training. The sample selection will follow the multi-center principle. The olfactory training (OT) intervention will last for 12 weeks.

Evaluation The primary endpoint will be the change in olfactory ability from baseline to the 12-week intervention or control period. The intervention effect will be evaluated by the total score of the Sniffer Stick Test (SST)-Threshold, Discrimination and Identification (TDI)-Extended Version. Secondary endpoints will be changes in olfactory bulb volume and shape, olfactory-related brain area volume, olfactory and trigeminal nerve-related potentials, and cognitive questionnaires.

Conclusion（objective） The present study aimed to explore the efficacy of the modified olfactory training device (MOT), and compare COT and MOT with respect to the resultant improvement in olfactory function.

At the same time, our study will use a variety of outcome indicators to evaluate the changes in patients before and after treatment, which will lay the foundation for exploring the mechanism of olfactory training in treating patients with post-viral olfactory disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, gender not limited.
2. Patients diagnosed with olfactory dysfunction following infections of the upper respiratory tract, as determined by Sniffin' Sticks test (including TDI value test).
3. Voluntarily signs the informed consent form.

Exclusion Criteria:

1. Patients with post-traumatic olfactory dysfunction, rhinosinusitis-related dysfunction and olfactory dysfunction caused by other reasons.
2. Patients with concomitant sinonasal disease.
3. Patients with chronic diseases, such as hypertension, diabetes, bronchopneumonia, chronic obstructive pulmonary disease, etc.
4. Patients with serious coexisting diseases: such as malignant tumors, etc., with a life expectancy of less than 2 years.
5. Patients who cannot tolerate olfactory function testing and treatment.
6. Patients who have taken oral glucocorticoids, antibacterial drugs, anti-leukotrienes, antihistamines, or received olfactory training within four weeks will be excluded.
7. Patients who are receiving treatment that affects olfactory recovery.
8. Patients with smoking habits.
9. Patients who are already or plan to be pregnant.
10. According to the judgment of the researchers, the patient cannot complete this study or cannot comply with the requirements of this study (such as memory or behavior abnormalities, depression, heavy drinking, previous breach of contract).
11. Patients who did not consent for participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-22 (Estimated); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
The total scores in the "Sniffin 'Sticks" test | Baseline,Month 3,Month 6,Month 12,Month 24
  This olfactory test consists of three subtests that respectively measure odor threshold (T), odor discrimination (D), and odor identification (I). Each subtest has a maximum score of 16, and the sum of the scores from the three subtests provides the global olfactory score (TDI score; Threshold, Discrimination, Identification) with a maximum of 48 points. Patients with a TDI composite score≥30.5 are defined as normosmic. In contrast, those with a TDI composite score between 16.5 and 30.5 are defined as hyposmic, and patients with a TDI composite score<16.5 are defined as functionally anosmic. Based on previous literature, we have established a 5.5 points improvement in the TDI composite score as a significant change.

SECONDARY OUTCOMES:
OB volume and shape measurement | Baseline,Month 3,Month 6,Month 12,Month 24
  OB volumetric evaluations will be performed with a 3-Tesla MRI system with coronal T2-weighted fast spin-echo images that included the anterior and the middle parts of the skull base.
  The OB volume will be measured using manual segmentation. The contours of the left and the right OBs will be manually delineated. The proximal limit of the OB will be determined on the basis of the sudden change in the diameter at the beginning of the olfactory tract. After all surfaces are added and multiplied by the slice thickness, the volume in cubic millimeters will be obtained for the right and the left OBs, and the total OB volume will be calculated as the sum of the two values.
  Measurements will be performed blindly twice by two examiners. When the difference in volume is > 10%, the examiners will perform a third measurement together.
  We have interpreted oval, round, triangular, and bean/boat/banana shapes as normal variants of OB shape.Atrophy will be interpreted as flattened OB.
MRI volumetric evaluation related to GM | Baseline,Month 3,Month 6,Month 12,Month 24
  Magnetic resonance imaging (MRI) scans will be performed on a 3T Siemens Verio scanner with a 12-channel phased-array head coil,measuring gray matter(GM) volumes to explore the connection between olfactory function and brain regions.
MRI volumetric evaluation related to WM | Baseline,Month 3,Month 6,Month 12,Month 24
  Magnetic resonance imaging (MRI) scans will be performed on a 3T Siemens Verio scanner with a 12-channel phased-array head coil,measuring white matter(WM) volumes to explore the connection between olfactory function and brain regions.
MRI volumetric evaluation related to CSF | Baseline,Month 3,Month 6,Month 12,Month 24
  Magnetic resonance imaging (MRI) scans will be performed on a 3T Siemens Verio scanner with a 12-channel phased-array head coil,measuring cerebrospinal fluid(CSF) volumes to explore the connection between olfactory function and brain regions.
Event-related potentials (ERPs) | Baseline,Month 3,Month 6,Month 12,Month 24
  Event-related potentials include olfactory event-related potentials(oERPs) and trigeminal event-related potentials (tERPs).
  We will use an OM6b olfactometer to generate ERPs after we have stimulated patients with phenethyl alcohol per standard methods.We infuse olfactory- and then trigeminal-nerve stimuli into the nasal cavity at a constant temperature and flow rate.We will place reference electrodes in the left and right earlobes When analyzing the records offline, we will exclude those contaminated by blinking or other interference . After amplification and filtering, we will obtain stable oERPs and tERPs waveforms.
Questionnaire of Olfactory Disorders | Baseline,Month 3,Month 6,Month 12,Month 24
  Questionnaire of Olfactory Disorders (QOD) determines the impact of olfactory dysfunction on daily life (70). The QOD consists of 52 statements, which can be divided into 3 domains: 39 negative statements (degree of suffering; NS), 5 positive statements (positive effects and coping strategies) and 8 socially desired statements ("lie scale") .
Visual analogue scale for olfactory training | Baseline,Month 3,Month 6,Month 12,Month 24
  Subjective ratings of olfactory function will be also recorded at baseline and follow-up appointments by means of a visual analogue scale, scoring from 0 to 100. On this scale, 0 represents complete olfactory loss and 100 perfect olfactory function. In addition, patients were asked about the presence of qualitative olfactory disorders such as parosmia.

CONTACTS AND LOCATIONS:
Locations (1):
- Bejing, Beijing, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.

REFERENCES:
- [Derived] Xie J, Li Y, He H, Liu Y, Chen L, Liu X, Zhao D, Wu D. Randomised trial protocol to assess efficacy of modified olfactory training method for patients with postinfectious olfactory dysfunction. BMJ Open. 2025 Dec 23;15(12):e101183. doi: 10.1136/bmjopen-2025-101183. PMID 41436263